CLINICAL TRIAL: NCT02970474
Title: A Study Utilizing 3D Printing in Patients Undergoing External Beam Radiation Therapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment and loss of co-investigator.
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-933857
Record Dates: First submitted 2016-11-18; First posted 2016-11-22 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Other): All participants will undergo the same schedule. Each participant will be fitted with a conventional and a 3D printed bolus prior to receiving radiation therapy. Each bolus will be assessed for optimal dose distribution of the radiation to the tumor through computer stimulation. The bolus, either conventional or 3D printed, that is found to be superior will be used for the actual radiation therapy treatment.
  Interventions: Device: Conventional Bolus; Device: 3D Printed Bolus

INTERVENTIONS:
Device: Conventional Bolus — Conventional bolus is mold made from Super stuff powder, superflab, or paraffin wax and made to fit the contours of the body.
Device: 3D Printed Bolus — The 3D printed bolus is also made from Super stuff powder, superflab, or paraffin wax, however it uses CT scans to print a molded bolus from the images of the participant's body.

SUMMARY:
Some radiation therapy treatment plans require the use of boluses. Boluses are placed directly on the skin overlying the area to be treated. The radiation beam interacts with the bolus before entering the body and ensures that the correct radiation dose reaches your tumor. The purpose of this study is to determine whether the shortcomings of conventional bolus preparation can be overcome by using a 3D printer. CT scans of the body can be used to create 3D models for boluses. The 3D models can then be printed into plastic boluses using a 3D printer. Preliminary studies have shown that 3D printed boluses conform to body contours better and allow for more precise control over radiation dose. In this study, both a conventional and 3D printed bolus will be made. The Investigators will then simulate treatment with both boluses to determine which bolus will result in more optimal treatment for the participant. The superior bolus will be used in the participant's treatment.

DETAILED DESCRIPTION:
In radiation therapy, high-energy radiation beams treat tumors by damaging cancer cells. Treatment plans are designed with the goal of limiting exposure to adjacent healthy tissues. Commonly used radiation beams demonstrate the "skin-sparing effect" which means that the radiation dose builds up after the beam enters the skin and thus the maximum dose is reached at some depth beneath the skin. For many tumors, this spares the skin from unnecessary exposure while ensuring cancer cells beneath the skin receive the maximum dose. For cancers that lie at or just below the skin surface, however, it is desirable for the maximum dose be present at the skin surface. In such cases, a bolus (material with properties similar to tissue) is used to mimic tissue and is placed above the skin. Dose build up occurs within the bolus, thus allowing the maximum dose to be reached at the skin surface. Aside from the treatment of superficial tumors, boluses have recently been used for modulated electron radiation therapy (MERT). For MERT, the bolus thickness is varied so that the dose at a specific depth can be varied at different locations within the tissue. With this technique, the bolus is customized for a patient's specific anatomy and thus radiation exposure to healthy tissue is minimized.

Boluses are typically made from moldable materials such as paraffin wax or superflab. Conventional bolus preparation has its disadvantages; the patient is required to be present, it can be time intensive and it is dependent on the skill of the fabricator. Furthermore, the degree of conformity to the patient's skin is limited and, as a result, there can be significant air gaps between the bolus and the patient's skin. Such air gaps have been shown to create significant reduction in the surface dose.

The goal of the present study is to improve the current process of bolus preparation by creating customized boluses with 3D printing. Customized boluses can be designed in Varian eclipse software and then imported into 3D modeling software such as 3D Slicer. The 3D model can then be converted into STL (Stereolithography) format which can be interpreted by the 3D printer software. Several preliminary studies have reported success in creating such boluses. One study reported good fit without air gaps (Kim) in their 3D printed bolus. Additionally, several studies modeled tissue dose distributions for 3D printed boluses and found results were similar to those obtained for conventional boluses.

For the current study, the Investigators will enroll participants who require boluses as part of their treatment plan. Both a conventional and 3D bolus will be fabricated for each participant. Computer simulation of dose distributions will be used to compare dosimetric parameters. Additionally, air gaps for both boluses will be measured. For each participant, the bolus that results in a more optimized dose distribution will be used for the participant's actual treatment. Conducting the study will necessitate each enrolled participant to undergo an additional CT scan to simulate treatment with the 3D printed bolus.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Requires bolus and is schedule for radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Optimal radiation dose | 1 day
  Boluses are used in radiation therapy to assure the optimal dose of radiation is applied to the tumor. Conventional boluses may have air gaps between the mold and the participants skin, or deform over time and use, which may make the dose of radiation change and not be at the optimal dose for the tumor. Therefore a 3D printed bolus will be molded based on a participant's CT images to construct a bolus to deliver the optimal dose of radiation to the tumor. Both boluses will be tested through a computer simulation to asses which bolus, conventional or 3D printed, provides the optimal radiation dose.

CONTACTS AND LOCATIONS:
Overall Officials: Steven DiBase, MD, Principal Investigator — Tulane University
Locations (1):
- Tulane University Cancer Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share IPD.